CLINICAL TRIAL: NCT04747483
Title: Effects of Extension Oriented Treatment Approach (EOTA) With Or Without Mechanical Traction For Patients With Lumbar Spondylosis
Brief Title: EOTA With Or Without Mechanical Traction For Patients With Lumbar Spondylosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00774 Aroosa Bibi
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Lumbar Spondylosis
Keywords: Lumbar Spondylosis, EOTA, Mechanical traction
MeSH Terms: conditions — Spondylosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extension Oriented Treatment Approach (Active Comparator): The EOTA intervention involves three components. The first component is a series of active extension- oriented exercises: Prone lying: Able to tolerate for 5 minutes, no pillow Prone lying on elbows: Able to tolerate for 5 minutes Prone press up exercise: 3 sets of 10 repetitions, move to end-range extension Repeated extension in standing: 3 sets of 10 repetitions, move to end-range extension.
  The second component of the EOTA is subject education. Subjects are being educated to maintain the natural lordosis of the lumbar spine while sitting, and are being instructed to avoid prolonged sitting for greater than 20-30 minutes whenever possible.
  The third component of the EOTA is mobilization of the lumbar spine to promote lumbar extension.The mobilization component consist of a series of up to 20 graded oscillatory mobilizations performed with the subject prone by using a grade I - IV mobilization force as described by Maitland.
  Interventions: Other: Extension Oriented Treatment Approach
- EOTA+ Mechanical Traction (Experimental): Subjects in the EOTA + traction group receive the EOTA components described above with Mechanical lumbar traction.
  Intermittent traction being applied (30-sec hold, 10-sec rest) for 15 minutes. Traction started with 25% of the patients' body weight and increased until the patient indicated that the tolerance for pulling was reached, with a maximum of 50% of the total body weight.
  2 sessions being given per week for 3 weeks.
  Interventions: Other: EOTA+ Traction

INTERVENTIONS:
Other: Extension Oriented Treatment Approach — The EOTA intervention involves three components.
  The first component is a series of active extension- oriented exercises:
  Prone lying: Able to tolerate for 5 minutes, no pillow Prone lying on elbows: Able to tolerate for 5 minutes Prone press up exercise: 3 sets of 10 repetitions, move to end-range extension Repeated extension in standing: 3 sets of 10 repetitions, move to end-range extension The second component of the EOTA is subject education. Subjects are educated to maintain the natural lordosis of the lumbar spine while sitting, and are instructed to avoid prolonged sitting for greater than 20-30 minutes whenever possible.
  The third component of the EOTA is mobilization of the lumbar spine to promote lumbar extension. The mobilization component consist of a series of up to 20 graded oscillatory mobilizations performed with the subject prone by using a grade I - IV mobilization force as described by Maitland.
  Other Names: EOTA
  Arms: Extension Oriented Treatment Approach
Other: EOTA+ Traction — Subjects in the EOTA + traction group receive the EOTA components described above with Mechanical lumbar traction.
  Intermittent traction being applied (30-sec hold, 10-sec rest) for 15 minutes. Traction started with 25% of the patients' body weight and increased until the patient indicated that the tolerance for pulling was reached, with a maximum of 50% of the total body weight.
  2 sessions being given per week for 3 weeks.
  Arms: EOTA+ Mechanical Traction

SUMMARY:
The aim of this research is to find and compare the effect of extension oriented treatment approach with or without mechanical traction on pain, range of motion and disability in patients with lumbar spondylosis. Randomized controlled trial is being conducted at Women Institute of Rehabilitation sciences. The sample size is 70. The subjects are being divided in two groups, 35 subjects in extension oriented treatment approach (EOTA) group and 35 in EOTA + traction group. Study duration is of 6 months. Sampling technique being applied is purposive non probability sampling technique.Tools being used in the study are Numeric pain rating scale (NPRS), Goniometer and Oswestry disability index (ODI).

DETAILED DESCRIPTION:
Lumbar spondylosis is a degenerative condition of lower lumbar spine that presents with chronic low back pain that last from more than three months and is aching in nature and radiates to lower limbs. Lumbar region pain, range of motion restriction and limitation in functions are features of lumbar spondylosis. Symptoms of lumbar spondylosis include low back pain, radicular pain, numbness of leg, weakness of leg and neurogenic claudication. Lumbar spine degenerative disorders are normal, age related phenomena. Repetitive loading of the spine, abnormal working postures and repeated movements can all lead to the degenerative changes in the spine. Low back pain due to degenerative changes disturb the individual functional activities. Mechanistically spondylosis is the hypertrophic response of adjoining vertebral bone to degenerative disk. The term spondylosis nonspecifically can be applied to degenerative changes affecting the discs and vertebral bodies and associated joints of the lumbar spine. Decrease in the height of disk lead to increase in loads on the facet joints.

In LBP rehabilitation the challenge is to arrive at any basic general rehabilitation care paradigms that would apply to most sub populations of low back. The goals of physical therapy management for patients with low back pain are to control pain, restore function and prevent future functional deficits.

Substantial variation in management by conservative and invasive approaches exists between practitioners throughout the country. Treatment options for the management of chronic low back pain syndromes include: physical therapy (and associated modalities and behavioral techniques), pharmacotherapy, injection therapy, and surgical intervention. Exercise therapy (ET) remains one of the conservative mainstays of treatment for chronic lumbar spine pain, and may be tailored to include aerobic exercise, muscle strengthening, and stretching exercises. TENS, Back School (concepts of posture, ergonomics, and appropriate back exercises), Lumbar back supports, traction and spine manipulation are other treatment methods commonly used for treating low back pain. Delito and colleagues described the treatment based classification system (TBC) is a classification approach for low back pain. The treatment based classification system includes subgroup of subjects with lumbar conditions that benefits from an Extension oriented treatment approach. EOTA includes active and passive activities combination to promote lumbar spine extension. EOTA exercises are used to reduce leg symptoms or promote centralization. Several studies provided evidence that subgrouping classification methods use for the physical therapist management of LBP patients provide better outcomes than physical therapy management that is not based on classification. Randomized controlled trials using TBC for patients with LBP of acute and sub-acute have reported significant outcomes compared with usual care or random interventions.

Lumbar traction is a popular modality used for patients with chronic LBP. Many healthcare and physical therapist utilized it for treating chronic LBP. Research suggests that certain LBP patients benefit from lumbar traction. Traction mechanical effects involve lordosis reduction, separating the facets, intervertebral foramen opening and eliminating muscles spasms. Pressure caused by gravity and soft tissues reduced by traction therapy, and adequate tension allows intervertebral disc, vertebra, and spinal nerves separation. It is suggested that elongation of spine inhibits nociceptive impulses by increases intervertebral space and reducing lumbar lordosis and also, releases adhesions around the zygapophysial joint and the annulus fibrosus and decreases mechanical stress. Evidence of Physiotherapy with traction versus physiotherapy without traction showed lower mean pain intensity in the traction group (a difference of 7.96 points on the VAS, 95% CI -16.53 to 0.61) at one to two weeks' follow-up.

Most previous studies have not examined effects of an EOTA with or without traction for patients with lumbar spondylosis. The purpose of this study is to examine the effects of an EOTA with or without traction for patients with lumbar spondylosis.

Sharma A, Alahmari K, Ahmed I conducted a research Efficacy of Manual Therapy versus Conventional Physical Therapy in Chronic Low Back Pain Due to Lumbar Spondylosis. Total of 30 samples of subjects were assigned into two groups in this study. Group -I received Maitland mobilization and lumbar stabilization exercises and group-II received conventional physical therapy (traction, strengthening, stretching exercises). Then outcomes were assessed. The results showed that managing low back pain, range of motion and function of the lumbar spine manual therapy interventions are more effective than conventional physical therapy.

Research by David A Browder, John D Childs, Joshua A Cleland, and Julie M Fritz which is the Effectiveness of an Extension-Oriented Treatment Approach in a Subgroup of Subjects with Low Back showed that the EOTA group demonstrated greater change in pain at the 1-week follow-up only. An EOTA was more effective than trunk strengthening exercise in a subgroup of subjects hypothesized to benefit from this treatment approach.

In a study by Anne Thackeray et al which is to examine the effectiveness of mechanical traction in patients with lumbar nerve root compression and within a predefined subgroup. In this study criteria of predefined subgrouping was used and patients were randomized to receive an extension oriented treatment approach with or without the mechanical traction addition. The results of this study concluded that there is no evidence that addition of lumbar mechanical traction with an extension oriented treatment is more beneficial to extension oriented treatment alone for the predefined subgroup of patient's management.

A case report by Allison R. Gagne & Scott M. Hasson (2010) Lumbar extension exercises in conjunction with mechanical traction for the management of a patient with a lumbar herniated disc. In this case report mechanical traction in addition with lumbar extension exercises was used for a patient with lumbar herniated disc and purpose was to describe and discuss its use. The results indicated that goals for the patient were achieved and the patient complaint of numbness and tingling was no more present. Patient improvement of pain and prior function level was achieved with lumbar extension exercises in addition with mechanical traction this case report data suggests.

ELIGIBILITY:
Inclusion Criteria:

- Mild to moderate level chronic low back pain with or without radiation of pain History of slow, insidious onset of pain from three months

On Physical examination:

* Limited ROMs of lumbar spine i.e. extension (< 20 degrees), flexion (< 40 degrees) or side flexion (< 15 degrees).
* Extension may be more limited than other movements.
* Pain during extension like standing and relieved by flexion like sitting.
* Pins and needles sensations (two out of over four should be there).
* Nature of pain-aching pain, feeling of heaviness in legs, intermittent burning or numbness.
* No neurological deficits.
* Diagnosis confirmed by X-Ray /MRI showing signs of degeneration.

Exclusion Criteria:

* Fractures
* Evidence of central nervous system involvement, including symptoms of cauda equina syndrome (i-e loss of bowl or bladder control) in the physical examination
* Recent (within the past 2 weeks) LBP
* Pregnancy
* Malignancy
* Spondylolisthesis
* Mechanical strain
* Previous back surgery
* Other red flags (contraindications to surgery)

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index: | Three weeks
  The ODI is a 10-item questionnaire designed to assess disability in typical daily activities. Scoring ranges from 0 to 100, with higher scores 100 indicating greater disability.

SECONDARY OUTCOMES:
NPRS | Three weeks
  Changes from base Line Numeric Pain rating scale is a scale for pain starting from 0-10. Where 0 indicate no pain and 10 indicate severe pain.

OTHER OUTCOMES:
ROM Lumbar Spine | three weeks
  Changes from the Baseline ROM range of Motion of Lumbar spine ROM being taken with the Help of Goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Asghar Khan, DScPT, Principal Investigator — Riphah International University
Locations (1):
- Women Institute of Rehabilitation Sciences, Abbottabad, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharma A, Alahmari K, Ahmed I. Efficacy of Manual Therapy versus Conventional Physical Therapy in Chronic Low Back Pain Due to Lumbar Spondylosis. A Pilot Study. Med Sci (Basel). 2015 Jun 26;3(3):55-63. doi: 10.3390/medsci3030055. PMID 29083391
- [Background] Saetia K, Kuonsongtham V. Central Spinal Canal Decompression for Lumbar Spondylosis with Uniportal Full-Endoscopic Interlaminar Approach: Technical Note and Preliminary Results in Thailand. J Med Assoc Thai. 2016 Jun;99 Suppl 3:S16-22. PMID 29901333
- [Background] George BA, Shinde SB. Effect of activity specific spinal stabilization exercises on pain and spinal mobility in lumbar spondylosis. Int J Health Sci Res. 2019; 9(7):174- 182.
- [Background] Middleton K, Fish DE. Lumbar spondylosis: clinical presentation and treatment approaches. Curr Rev Musculoskelet Med. 2009 Jun;2(2):94-104. doi: 10.1007/s12178-009-9051-x. Epub 2009 Mar 25. PMID 19468872
- [Background] Uduonu E. Cardiopulmonary adaptation to 6- weeks' skin traction and isometric exercise among Nigerian subjects with lumber spondylosis 2017.
- [Background] Pergolizzi JV Jr, LeQuang JA. Rehabilitation for Low Back Pain: A Narrative Review for Managing Pain and Improving Function in Acute and Chronic Conditions. Pain Ther. 2020 Jun;9(1):83-96. doi: 10.1007/s40122-020-00149-5. Epub 2020 Jan 31. PMID 32006236
- [Background] Browder DA, Childs JD, Cleland JA, Fritz JM. Effectiveness of an extension-oriented treatment approach in a subgroup of subjects with low back pain: a randomized clinical trial. Phys Ther. 2007 Dec;87(12):1608-18; discussion 1577-9. doi: 10.2522/ptj.20060297. Epub 2007 Sep 25. PMID 17895350
- [Background] Ojha H, Egan W, Crane P. The addition of manipulation to an extension-oriented intervention for a patient with chronic LBP. J Man Manip Ther. 2013 Feb;21(1):40-7. doi: 10.1179/2042618612Y.0000000014. PMID 24421612
- [Background] Tadano S, Tanabe H, Arai S, Fujino K, Doi T, Akai M. Lumbar mechanical traction: a biomechanical assessment of change at the lumbar spine. BMC Musculoskelet Disord. 2019 Apr 9;20(1):155. doi: 10.1186/s12891-019-2545-9. PMID 30961554
- [Background] GŬLŞEN, MUSTAFA, et al.
- [Background] Bilgilisoy Filiz M, Kilic Z, Uckun A, Cakir T, Koldas Dogan S, Toraman NF. Mechanical Traction for Lumbar Radicular Pain: Supine or Prone? A Randomized Controlled Trial. Am J Phys Med Rehabil. 2018 Jun;97(6):433-439. doi: 10.1097/PHM.0000000000000892. PMID 29309314
- [Background] Ozturk B, Gunduz OH, Ozoran K, Bostanoglu S. Effect of continuous lumbar traction on the size of herniated disc material in lumbar disc herniation. Rheumatol Int. 2006 May;26(7):622-6. doi: 10.1007/s00296-005-0035-x. Epub 2005 Oct 25. PMID 16249899
- [Background] Fritz JM, Thackeray A, Childs JD, Brennan GP. A randomized clinical trial of the effectiveness of mechanical traction for sub-groups of patients with low back pain: study methods and rationale. BMC Musculoskelet Disord. 2010 Apr 30;11:81. doi: 10.1186/1471-2474-11-81. PMID 20433733
- [Background] Gagne AR, Hasson SM. Lumbar extension exercises in conjunction with mechanical traction for the management of a patient with a lumbar herniated disc. Physiother Theory Pract. 2010 May;26(4):256-66. doi: 10.3109/09593980903051495. PMID 20397860